CLINICAL TRIAL: NCT06864572
Title: Clinical Application of Dual-target Imaging Agent [68Ga]Ga-P17-079 in the Diagnosis and Treatment of Metastatic Prostate Cancer
Brief Title: [68Ga]Ga-P17-079 in the Diagnosis and Treatment of Metastatic Prostate Cancer
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-NM-079
Record Dates: First submitted 2025-02-19; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Prostate Cancer (mPC)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- P17-079+P16-093 (Experimental)
  Interventions: Diagnostic Test: P17-079, P16-093, or P15-041 PET/CT
- P17-079+P15-041 (Experimental)
  Interventions: Diagnostic Test: P17-079, P16-093, or P15-041 PET/CT

INTERVENTIONS:
Diagnostic Test: P17-079, P16-093, or P15-041 PET/CT — P17-079, P16-093, or P15-041 PET/CT

SUMMARY:
Preclinical studies have confirmed that [68Ga]Ga-P17-079 in both mouse prostate tumors and osseogenic metastases has high uptake and prolonged retention, which enables [68Ga]Ga-P17-079 to be fully absorbed by the lesions, and it is possible to detect bone metastases, prostate cancer primary sites, lymph node metastases and organ metastases at the same time in a single examination. It is a potential "killing two birds with one stone" imaging agent. At this stage, the clinical study of [68Ga]Ga-P17-079 in the diagnosis and treatment of metastatic prostate cancer as a self-made preparation is planned to be carried out in our hospital to further verify its clinical application value.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18-85 years, expected survival ≥12 weeks.
* Patients who have not undergone chemoradiotherapy, feasible surgery or biopsy to obtain a pathological diagnosis or are highly suspected of malignancy according to clinical diagnostic criteria.
* At least one measurable target lesion was present according to RECIST1.1 criteria.
* Obtain written informed consent and be able to follow up

Exclusion Criteria:

* Severe abnormal liver and kidney function
* Fertile subjects will need to use effective contraception during the study
* Unable to lie flat for half an hour
* Refused to join this clinical investigator
* Suffering from claustrophobia or other mental illness
* Other conditions deemed unsuitable for participation in the trial

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
SUV | 0-180 min post-injection
  measured by PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided